CLINICAL TRIAL: NCT06731387
Title: Impact of Implementing Pharmaceutical Technical Assistants to Support the Medication Process in Hospital Wards: Effects on Operational Efficiency and Medication Safety
Brief Title: Assessing the Role of Pharmaceutical Technical Assistents in Hospital Wards: Measuring Efficiency and Medication Safety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaz (Other)
Collaborators: Universiteit Antwerpen (Other); University of Applied Sciences Utrecht (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EC24018
Record Dates: First submitted 2024-12-02; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Medication Safety; Time Efficiency; Interdepartmental Communication
Keywords: pharmacy assistants; medication safety; hospital ward; medication management; nursing

STUDY DESIGN:
Intervention Model Description: This study focuses on analyzing 50 medication dispensation processes on hospital wards, evenly distributed across two distinct periods: a control period without the involvement of Pharmaceutical Technical Assistants (PTAs) (medication dispensation by the night nurses) and an intervention period where PTAs actively participate in medication dispensation. Nurses and PTAs observed during the dispensation processes will be included in the study based on the selected medication dispensation moments during which they are on duty.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PTAs dispensing medications (Experimental)
  Interventions: Other: Pharmaceutical technical assistants supported medication dispensation on the hospital ward

INTERVENTIONS:
Other: Pharmaceutical technical assistants supported medication dispensation on the hospital ward — Pharmaceutical technical assistants (PTAs) visit the hospital ward for two hours in the morning or afternoon to dispense medications for admitted patients for the following day. Night nurses then complete any final additions or adjustments as needed.

SUMMARY:
The goal of this interventional study is to evaluate the impact of implementing pharmaceutical technical assistants (PTAs) to support the medication process on hospital wards on operational efficiency and medication safety among nurses and pharmaceutical technicial assistants. The main questions it aims to answer are:

* What is the effect of PTAs on the time spent by (night) nurses on medication dispensation?
* How does their involvement influence unplanned interactions between nursing staff and the pharmacy?
* What is the impact of PTAs on the safety of medication processes, including missed or delayed doses, accuracy of dispensed medication, and reported medication errors?

Researchers will compare periods with and without the involvement of PTAs in the medication management process on the hospital ward to assess differences in:

* Time spent on medication dispensation.
* Frequency of unplanned interactions between hospital wards and the pharmacy.
* Rates of missed or delayed medication doses.
* Accuracy of dispensed medication compared to prescriptions.
* Reported medication errors.

During the observed medication dispensation processes, involved nurses and PTAs will:

* Be observed while preparing medications to measure time and interruptions.
* Provide data on medication errors and delays through digital systems and reports.
* Complete a demographic questionnaire about their professional background. This study involves both intervention and control periods, allowing researchers to measure the specific effects of PTAs' involvement in medication processes.

ELIGIBILITY:
Inclusion Criteria for observed medication dispensation moments

Control Period:

* Medication dispensation moments must be performed by nurses during the nightshift. .
* Nurses included must have at least six months of experience working night shifts.

Intervention Period:

* Medication dispensation moments must be performed by PTAs.
* PTAs included must have at least six months of experience specifically in medication dispensation tasks.

Exclusion Criteria: Hospital wards that introduced the involvement of PTAs less than six months ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Time spent on medication dispensation on the hospital ward | Data collection was conducted over five days during the control period and five days during the intervention period on each of the included hospital wards.
  Intervention Period:
  Observing and recording the time the Pharmaceutical Technical Assistant (PTA) spends dispensing medication on the hospital ward.
  This is followed by observing and recording the time the night nurse takes to complete the medication dispensation for the next day.
  Control Period:
  Observing and recording the time the night nurse spends dispensing medication for the next day without PTA involvement.

SECONDARY OUTCOMES:
Dispensing errors | Data collection was conducted over five days during the control period and five days during the intervention period on each of the included hospital wards.
  Intervention Period: Verifying the accuracy of medication dispensed by the PTA, including recording the number and type of errors identified.
  Control Period: Verifying the accuracy of medication dispensed by the night nurse, including recording the number and type of errors identified.
Delayed and omitted medication doses | Data collection was conducted over five days during the control period and five days during the intervention period on each of the included hospital wards.
  Intervention Period:
  Reviewing the electronic medication system for the day the PTA prepared the medication. This includes recording the number of delayed or missed doses, the name and type of medication involved, and the reasons for the delay or non-administration.
  Control Period:
  Reviewing the electronic medication system for the day the night nurse dispensed the medication. This includes recording the number of delayed or missed doses, the name and type of medication involved, and the reasons for the delay or non-administration.
Reported Medication Errors | Data collection was conducted over five days during the control period and five days during the intervention period on each of the included hospital wards.
  Collecting the reported medication errors from the hospital's incident reporting system during both the intervention and control periods.
Interdepartmental Communication Between Pharmacy and Hospital Ward | Data collection was conducted over five days during the control period and five days during the intervention period on each of the included hospital wards.
  The exchange of information and updates between the pharmacy and the hospital ward to ensure accurate medication preparation, timely delivery, and proper administration. During both the intervention and control periods, this communication includes coordinating medication orders, addressing discrepancies, managing urgent requests, and providing guidance or clarifications as required.

CONTACTS AND LOCATIONS:
Overall Officials: Tinne Dilles, Doctor, Professor, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Vitaz, Sint-Niklaas, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rathbone AP, Jamie K, Blackburn J, Gray W, Baqir W, Henderson E, Campbell D. Exploring an extended role for pharmacy assistants on inpatient wards in UK hospitals: using mixed methods to develop the role of medicines assistants. Eur J Hosp Pharm. 2020 Mar;27(2):78-83. doi: 10.1136/ejhpharm-2018-001518. Epub 2018 Sep 3. PMID 32133133
- [Background] Kjeldsen LJ, Schlunsen M, Meijers A, Hansen S, Christensen C, Bender T, Ratajczyk B. Medication Dispensing by Pharmacy Technicians Improves Efficiency and Patient Safety at a Geriatric Ward at a Danish Hospital: A Pilot Study. Pharmacy (Basel). 2023 May 8;11(3):82. doi: 10.3390/pharmacy11030082. PMID 37218964